CLINICAL TRIAL: NCT03004209
Title: Effect of Erythropoietin in Refractory Autoimmune Encephalitis Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607-120-777
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Autoimmune Encephalitis
Keywords: Erythropoietin; Autoimmune encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EPO (Other): Erythropoietin injection: three times per a week, 100 IU/kg for each patients Trade name: epokine prefilled injection
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — three times per a week 100IU / k
  Other Names: Epokine prefilled injection

SUMMARY:
This study evaluates the efficacy of erythropoietin in refractory autoimmune encephalitis. Ten patients will receive 100 IU/kg of erythropoietin 3 times a week for 12 weeks.

DETAILED DESCRIPTION:
Erythropoietin can improve the refractory autoimmune encephalitis. Erythropoietin has tissue-protective effect via activation of Janus kinase (JAK)-2, signal transducer and activator of transcription (STAT)-5 pathway and NF-kappa B pathway. The activation of JAK-2 and STAT-5 promote hemoglobin synthesis and facilitate cell cycle progression. Also, NF-kappa B pathway inhibition regulates pro-inflammatory cytokine production.

We expect that erythropoietin may lead to improve the symptoms and outcome of autoimmune encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed autoimmune encephalitis
* Ineffective 1st line treatment (e.g. steroid IV, IVIg) and 2nd line treatment (e.g. Rituximab or cyclophosphamide)

Exclusion Criteria:

* Hemoglobin > 12g/dL
* Hematochrit >36%
* Thrombocytosis > 750K
* AST or ALT > 120
* HIV (+)
* Allergic reaction upon erythropoietin
* Uncontrolled hypertension
* mRS before the autoimmune encephalitis > 3
* Breast feeding or pregnancy
* History of ischemic stroke or pulmonary thrombosis
* Refuse to be enrolled

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline modified Rankin Scale (mRS) at 12th week | 2nd week, 12th week
  Favorable outcome is an improvement of mRS score.

SECONDARY OUTCOMES:
Adverse effect | 2nd week, 4th week, 8th week, 12th week
  Common terminology criteria for adverse events (CTCAE) 4.0
Quality of Life in Epilepsy Inventory (QOLIE) -31 | 2nd week, 4th week, 8th week, 12th week
Mini-Mental State Examination (MMSE) | 2nd week, 4th week, 8th week, 12th week

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No